CLINICAL TRIAL: NCT06349603
Title: Integrated Physiotherapy Approach for Susac Syndrome: A Comprehensive Case Study
Brief Title: Physiotherapy Approach for Susac Syndrome
Status: Completed | Type: Observational
Sponsor: Rehabilitation Centre Zivot (Other)
Responsible Party: Principal Investigator, Darko Bilic, Director, Rehabilitation Centre Zivot
Other Study IDs: S2023
Record Dates: First submitted 2024-03-29; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Susac Syndrome
Keywords: Physiotherapy
MeSH Terms: conditions — Susac Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Susac's syndrome is a rare autoimmune disorder characterised by a triad of encephalopathy (brain dysfunction), branch retinal artery occlusion (loss of vision) and sensorineural hearing loss. This study presents the case of a patient undergoing intensive physiotherapy intervention following an injury, focusing on assessments such as volume and range of motion measurements, manual muscle tests, and pain intensity evaluations using various scales.

DETAILED DESCRIPTION:
The patient, aged 17, initially presented with severe limitations in mobility, diagnosed with Susac syndrome. Requiring assistance to walk even short distances due to fear and insecurity. Through a structured physiotherapy program spanning several months, various assessments were conducted, including manual muscle tests and circumference measurements. Significant improvements were observed for muscle function, upper and lower limb circumferences, and performance in mobility tests.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Susac syndrome.
* Willingness and ability to participate in a 12-week intensive physiotherapy program.
* Stable medical condition that allows participation in physiotherapy without significant risks.
* Ability to provide informed consent for participation in the study.

Exclusion Criteria:

* Presence of severe comorbidities or medical conditions that would interfere with participation in physiotherapy or confound the study outcomes.
* Inability to comprehend or follow the instructions for physiotherapy exercises.
* Pregnancy, as certain physiotherapy modalities may not be suitable during pregnancy.
* Any other condition or circumstance that, in the opinion of the investigator, would compromise the safety or validity of participation in the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of a single adolescent patient diagnosed with Susac syndrome, aged 17 years. The patient presented with motor impairments and functional limitations attributed to Susac syndrome, including difficulties in mobility and muscle weakness. No significant comorbidities were reported, and the patient was medically stable to participate in a 12-week intensive physiotherapy program. Informed consent was obtained from the participant and their legal guardian prior to enrollment in the study."
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Mobility and Muscle Strength Improvement | Assessed at baseline and after 12 weeks of intensive therapy.
  This outcome measure evaluates improvements in mobility in a single individual with Susac syndrome following 12 weeks of intensive physiotherapy. Assessments include the Timed Up and Go test (TUG), which measures the time taken for the individual to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Progress is indicated by the transition from heavy reliance on assistance for mobility to independent walking for 100 meters.
Muscle Strength Improvement Outcome Measure | Assessed at baseline and after 12 weeks of intensive therapy.
  This outcome measure evaluates improvements in muscle strength in a single individual with Susac syndrome following 12 weeks of intensive physiotherapy. Assessments include manual muscle tests (MMT) to assess the strength and function of specific muscle groups, using a standardized grading scale. Progress is indicated by higher grades in manual muscle tests, reflecting improved muscle strength and endurance.
Pain Intensity Outcome Measure | Assessed at baseline and after 12 weeks of intensive therapy.
  This outcome measure evaluates changes in pain intensity experienced by the individual with Susac syndrome following 12 weeks of intensive physiotherapy. Pain intensity is assessed using the Visual Analog Scale (VAS), where the individual rates their pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain. Progress is indicated by a decrease in VAS scores, reflecting reduced pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation centre Život, Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmad A, Tariq F, Zaheer M. Incomplete Susac's Syndrome: A Case Report and Literature Review. Cureus. 2022 Aug 11;14(8):e27903. doi: 10.7759/cureus.27903. eCollection 2022 Aug. PMID 36110471
- [Background] Bose S, Papathanasiou A, Karkhanis S, Appleton JP, King D, Batra R, Mollan SP, Jacob S. Susac syndrome: neurological update (clinical features, long-term observational follow-up and management of sixteen patients). J Neurol. 2023 Dec;270(12):6193-6206. doi: 10.1007/s00415-023-11891-z. Epub 2023 Aug 22. PMID 37608221
- [Background] Coulette S, Lecler A, Saragoussi E, Zuber K, Savatovsky J, Deschamps R, Gout O, Sabben C, Aboab J, Affortit A, Charbonneau F, Obadia M. Diagnosis and Prediction of Relapses in Susac Syndrome: A New Use for MR Postcontrast FLAIR Leptomeningeal Enhancement. AJNR Am J Neuroradiol. 2019 Jul;40(7):1184-1190. doi: 10.3174/ajnr.A6103. Epub 2019 Jun 27. PMID 31248864
- [Background] Cvikova M, Stefela J, Vsiansky V, Dufek M, Dolezalova I, Vinklarek J, Herzig R, Zemanova M, Cervenak V, Brichta J, Barkova V, Kouril D, Aulicky P, Filip P, Weiss V. Case report: Susac syndrome-two ends of the spectrum, single center case reports and review of the literature. Front Neurol. 2024 Feb 16;15:1339438. doi: 10.3389/fneur.2024.1339438. eCollection 2024. PMID 38434197
- [Background] David C, Sacre K, Henri-Feugeas MC, Klein I, Doan S, Cohen FA, Jouvent E, Papo T. Susac syndrome: A scoping review. Autoimmun Rev. 2022 Jun;21(6):103097. doi: 10.1016/j.autrev.2022.103097. Epub 2022 Apr 10. PMID 35413469
- [Background] Egan RA. Diagnostic Criteria and Treatment Algorithm for Susac Syndrome. J Neuroophthalmol. 2019 Mar;39(1):60-67. doi: 10.1097/WNO.0000000000000677. PMID 29933288
- [Background] Luan X, Tian X, Zhang H, Huang R, Li N, Chen P, Wang R. Exercise as a prescription for patients with various diseases. J Sport Health Sci. 2019 Sep;8(5):422-441. doi: 10.1016/j.jshs.2019.04.002. Epub 2019 Apr 18. PMID 31534817
- [Background] Masjuan M, Ivanovski T, Sarasibar Ezcurra H, Rigo Oliver E. Behavioral Impairment and Amnesia at the Onset of Susac Syndrome. Cureus. 2023 Apr 25;15(4):e38089. doi: 10.7759/cureus.38089. eCollection 2023 Apr. PMID 37252530
- [Background] Patil S, Gs V, Sarode GS, Sarode SC, Khurayzi TA, Mohamed Beshir SE, Gadbail AR, Gondivkar S. Exploring the role of immunotherapeutic drugs in autoimmune diseases: A comprehensive review. J Oral Biol Craniofac Res. 2021 Apr-Jun;11(2):291-296. doi: 10.1016/j.jobcr.2021.02.009. Epub 2021 Feb 23. PMID 33948430
- [Background] Pereira S, Vieira B, Maio T, Moreira J, Sampaio F. Susac's Syndrome: An Updated Review. Neuroophthalmology. 2020 May 1;44(6):355-360. doi: 10.1080/01658107.2020.1748062. eCollection 2020. PMID 33408428
- [Background] Reedy MB, Wang Y, Beinlich BR, Rose WN. Successful Treatment of Incomplete Susac Syndrome with Simultaneous Corticosteroids and Plasmapheresis Followed by Rituximab. Case Rep Neurol Med. 2021 Aug 12;2021:5591559. doi: 10.1155/2021/5591559. eCollection 2021. PMID 34567813
- [Background] Rennebohm RM, Asdaghi N, Srivastava S, Gertner E. Guidelines for treatment of Susac syndrome - An update. Int J Stroke. 2020 Jul;15(5):484-494. doi: 10.1177/1747493017751737. Epub 2018 Jan 10. PMID 29319463
- [Background] Sveinsson O, Kolloch J, Traisk F, Brundin L. [Susac syndrome - an unusual syndrome which can be mistaken for multiple sclerosis]. Lakartidningen. 2020 Feb 10;117:FSSS. Swedish. PMID 32045006
- [Background] Wilf-Yarkoni A, Elkayam O, Aizenstein O, Oron Y, Furer V, Zur D, Goldstein M, Barequet D, Hallevi H, Karni A, Habot-Wilner Z, Regev K. Increased incidence of Susac syndrome: a case series study. BMC Neurol. 2020 Sep 2;20(1):332. doi: 10.1186/s12883-020-01892-0. PMID 32878610
- See also: Susac Syndrome: Collaboration is Required for a Diagnosis — https://clinmedjournals.org/articles/cmrcr/clinical-medical-reviews-and-case-reports-cmrcr-9-396.php?jid=cmrcr
- See also: Physiopedia contributors. (2022). Timed Up and Go Test (TUG). Physiopedia. — https://www.physio-pedia.com/Timed_Up_and_Go_Test_(TUG)
- See also: Physiopedia contributors. (2023). Benefits of Rehabilitation. Physiopedia. — https://www.physio-pedia.com/Benefits_of_Rehabilitation
- See also: Physiopedia contributors. (2024a). Assessing Range of Motion. Physiopedia. — https://www.physio-pedia.com/Assessing_Range_of_Motion
- See also: A case of possible Susac syndrome with avascular necrosis of hip — https://wjarr.com/sites/default/files/WJARR-2023-0294.pdf